CLINICAL TRIAL: NCT01451801
Title: Cellular Immunity in Adult Hepatitis B-vaccinated Serologic Non-responders
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Monash Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SJF0001
Record Dates: First submitted 2011-10-10; First posted 2011-10-14 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2012-10

CONDITIONS: Hepatitis B
Keywords: Hepatitis B; non responders; cellular immune response; cytokines; predictors; HBsAg
MeSH Terms: conditions — Hepatitis B | interventions — twinrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HBsAg (Other)
  Interventions: Biological: Twinrix

INTERVENTIONS:
Biological: Twinrix — A total of 400 healthy volunteers receive a standard course of immunization with a combined hepatitis A and B vaccine (Twinrix®) at 0, 1, and 6 months.
  Twinrix ® Adult suspension for injection. 1 ml contains 720 ELISA units of hepatitis A virus antigen adsorbed to aluminum hydroxide and 20 micrograms hepatitis B surface antigen (HBsAg) adsorbed to aluminum phosphate in sterile water. Excipient: sodium chloride. Contains traces of neomycin.

SUMMARY:
Previous studies have shown that 5-10% of Hepatitis B Virus vaccine recipients produce none or to few antibodies after a standard immunization with 3 vaccines. These individuals are defined as non-responders. The investigators wish to investigate if mounting another kind of immune response, called the cellular immune (CMI) response, protects these non-responders.

Aim/Hypothesis

Primary aims:

1. To estimate the CMI response in serologic non-responders after receiving a standard course of HBV immunization

   Secondary aims:
2. To establish the prevalence of serological non-responders after a standard course of HBV vaccination.
3. To assess the safety of the vaccine.
4. Evaluate predictors of serologic non-response in young, healthy individuals receiving a standard course of HBV immunization
5. To compare the immunological profile before and after a standard HBV vaccination regimen on non-responders and responders
6. Establish a rapid test for measuring CMI after being HBV vaccinated.

A total of 400 healthy volunteers receive a standard course of immunization with a combined hepatitis A and B vaccine (Twinrix®) at 0, 1, and 6 months. Blood is drawn at 0 and 8 months from all participants. The blood will be analysed to see if there is antibodies or/and if there is mounted a cellular immune response by measuring on parameters called cytokines.

ELIGIBILITY:
Inclusion Criteria:

* Signed participant information and consent
* Age over 18 years
* Women of childbearing potential must use effective contraceptives

Exclusion Criteria:

* previous HBV infection
* previous HBV immunization
* pregnancy (or planned pregnancy within 6 months)
* allergy to contents in the vaccine (formaldehyde).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Estimate the CMI response in serologic non-responders after receiving a standard course of HBV immunization | within 9. month from 1. vaccination
  Preparation of peripheral blood mononuclear cells (PBMC) Optimisation of antigen-specific cytokine flow cytometry Quantification of IFN-γ producing CD4+ T cells

SECONDARY OUTCOMES:
Establish the prevalence of serological non-responders after a standard course of HBV vaccination defined by anti-HBs <10 mIU / ml | Within 9 month from 1. vaccination
  Antibodies to Hepatitis B surface antigen are detected by use of a comercially available kit at the department of Clinical Immunology, Aarhus University Hospital, Skejby
Assess the safety of the vaccine by evaluating the numbers and intensity of adverse and Serious adverse events | Within 9 month from 1. vaccination
  By evaluating adverse events described in Case Report Forms
Evaluate predictors of serologic non-response in young, healthy individuals receiving a standard course of HBV immunization | within 9 month from 1. vaccination
  Questionnaire and *Magnitude of HBsAg-specific cell-mediated immune response.The presence of antigen specifik single, double or triple cytokine-producing T cells. Numbers and fractions of antigen-specific CD4 and CD8 T cells *HBsAg-specific T cell proliferation is quantified*The difference in phenotypic T cell profiles is getting compared at baseline*HBsAg-specific B cells measured by flow cytometry with staining for surface markers*Supernatant from HBsAg-stimulated PBMC is analysed regarding cytokines* Production of pro- og antiinflammatory cytokines is assesed by RT-PCR .
Compare the immunological profile before and after a standard HBV vaccination regimen, with com-parison of serological non-responders and serological responders | Within 9. month from 1. vaccination
  Magnitude of HBsAg-specific cell-mediated immune response.The presence of antigen specifik single, double or triple cytokine-producing T cells. Numbers and fractions of antigen-specific CD4 and CD8 T cells *HBsAg-specific T cell proliferation is quantified*The difference in phenotypic T cell profiles is getting compared at baseline*HBsAg-specific B cells measured by flow cytometry with staining for surface markers*Supernatant from HBsAg-stimulated PBMC is analysed regarding cytokines* Production of pro- og antiinflammatory cytokines is assesed by RT-PCR .
Establish a rapid test for measuring HBsAg specific CMI by use of an IFN-gamma based assay. | 18 month after 1. vaccination
  Preparation of peripheral blood mononuclear cells (PBMC) Optimisation of antigen-specific cytokine flow cytometry Quantification of IFN-γ producing CD4+ T cells

CONTACTS AND LOCATIONS:
Overall Officials: Lars Østergaard, Head, Study Chair — Department of Infectious Diseases, Aarhus University Hospital; Søren Jensen-Fangel, MD, Study Director — Department of Infectious Diseases, Aarhus University Hospital; Martin Tolstrup, MSc, Study Director — Department of Infectious Diseases, Aarhus University Hospital; Maria B Pedersen, Bach.Med, Principal Investigator — Department of Infectious Diseases, Aarhus University Hospital
Locations (1):
- Department of Infectious Diseases, Aarhus University Hospital, Aarhus N, Denmark